CLINICAL TRIAL: NCT03221920
Title: Effect of Very Low Carbohydrate Diet to Glasgow Prognostic Score, Serum Lactate and TNF Alpha on Colorectal Cancer Patients With Best Supportive Care
Brief Title: Very Low Carbohydrate Diet Effects to GPS, Serum Lactate and TNF Alpha on Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Soetomo General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DrSoetomoGH
Record Dates: First submitted 2017-07-16; First posted 2017-07-19 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Diet Modification; Colorectal Adenocarcinoma; Systemic Inflammation; TNF Alpha; Lactate
Keywords: Very Low Carbohydrate Diet; Colorectal Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Patients were randomized in to two groups, with very low carbohydrate diet and with normal diet
Who Masked: Care Provider
Masking Description: Care provider are not told whether the patient belongs to intervention or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very Low Carbohydrate Diet (Experimental): The patient will be evaluated for baseline clinical and laboratory values, and counselled on very low carbohydrate diet.
  Interventions: Other: Very Low Carbohydrate Diet
- Control (No Intervention): The patient will be evaluated for baseline clinical and laboratory values, and counselled on normal healthy .

INTERVENTIONS:
Other: Very Low Carbohydrate Diet — 1 : 4 ratio of carbohydrate to fat of the total daily calories intake
  Arms: Very Low Carbohydrate Diet

SUMMARY:
This study examine the effects of very low carbohydrate diet (in which the calories requirements are mostly from fat) to the level of systemic inflammation (measured by Glasgow Prognostic Score), serum lactate and TNF Alpha levels

DETAILED DESCRIPTION:
This study examine the effects of very low carbohydrate diet (in which the calories requirements are mostly from fat) to the level of systemic inflammation (measured by Glasgow Prognostic Score), serum lactate and TNF Alpha levels. The subjects are colorectal adenocarcinoma patients who were decided by experts to be managed by best supportive care. These patients are not deemed to be suitable for surgical intervention , chemotherapy or radiotherapy anymore. The main treatment is supportive. We would like to examined the effect of very low carbohydrate diet on these patients, in which theoretically tumtor cells of the colorectal adenocarcinoma needed glucose to replicate and increases the systemic inflammation response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as colorectal adenocarcinoma pathologically
* Decided by a digestive surgery consultant to be managed with best supportive care
* More than 17 years old and capable of making informed consent
* Karnofsky score > 50% or ECOG performance status <=2
* No clinical signs of infection, with one or more of these criteria : fever, leukocytosis, local sign of infection (eg.abscess,ulcer)
* AST < 2 times normal limit
* ALT < 2 times normal limit
* Serum Creatinine < 1,5 times normal limit
* Not pregnant (for women)
* Able to understand and willing participate and to sign informed consent form
* No Diabetes Mellitus
* No fat intolerance
* No severe malnutrition or cancer cachexia

Exclusion Criteria:

* Patient is still on other therapy for the tumour
* Patient with coexisting diseases which prohibits the patient to follow the study protocols

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2017-08-05 (Estimated); Primary Completion 2017-08-30 (Estimated); Study Completion 2017-08-30 (Estimated)

PRIMARY OUTCOMES:
Glasgow Prognostic Score | Change of baseline Glasgow Prognostic Score on day 21
  A score to evaluate systemic inflammation response

SECONDARY OUTCOMES:
Serum Lactate | Change of baseline Serum Lactate on day 21
  Lactate level in blood serum
TNF Alpha | Change of baseline TNF Alpha serum level on day 21
  Level of Tumor Necrosis Factor Alpha in the blood serum

CONTACTS AND LOCATIONS:
Overall Officials: Vicky S Budipramana, PhD, Principal Investigator — RS Dr Sutomo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sethi G, Sung B, Aggarwal BB. TNF: a master switch for inflammation to cancer. Front Biosci. 2008 May 1;13:5094-107. doi: 10.2741/3066. PMID 18508572
- [Background] Allen BG, Bhatia SK, Anderson CM, Eichenberger-Gilmore JM, Sibenaller ZA, Mapuskar KA, Schoenfeld JD, Buatti JM, Spitz DR, Fath MA. Ketogenic diets as an adjuvant cancer therapy: History and potential mechanism. Redox Biol. 2014;2:963-70. doi: 10.1016/j.redox.2014.08.002. Epub 2014 Aug 7. PMID 25460731
- [Background] Walenta S, Voelxen NF, Mueller-Klieser W. Lactate-An Integrative Mirror of Cancer Metabolism. Recent Results Cancer Res. 2016;207:23-37. doi: 10.1007/978-3-319-42118-6_2. PMID 27557533
- [Background] San-Millan I, Brooks GA. Reexamining cancer metabolism: lactate production for carcinogenesis could be the purpose and explanation of the Warburg Effect. Carcinogenesis. 2017 Feb 1;38(2):119-133. doi: 10.1093/carcin/bgw127. PMID 27993896
- [Background] Lasry A, Zinger A, Ben-Neriah Y. Inflammatory networks underlying colorectal cancer. Nat Immunol. 2016 Mar;17(3):230-40. doi: 10.1038/ni.3384. PMID 26882261
- [Background] Seyfried TN, Flores RE, Poff AM, D'Agostino DP. Cancer as a metabolic disease: implications for novel therapeutics. Carcinogenesis. 2014 Mar;35(3):515-27. doi: 10.1093/carcin/bgt480. Epub 2013 Dec 16. PMID 24343361
- [Background] Venetsanou K, Kaldis V, Kouzanidis N, Papazacharias Ch, Paraskevopoulos J, Baltopoulos G. Measurement of tumour necrosis factor receptors for immune response in colon cancer patients. Clin Exp Med. 2012 Dec;12(4):225-31. doi: 10.1007/s10238-011-0162-5. Epub 2011 Nov 1. PMID 22042432